CLINICAL TRIAL: NCT05480826
Title: Familial and Functional Study of Genetic Variants Identified in People With Schizophrenia, Bipolar Disorder, Autism Spectrum Disorder or Resistant Depression
Acronym: GENI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation FondaMental (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FF21-GENI; 2021-A02551-40 (Other: French National Agency for the Safety of Medicines and Health Products)
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: 2 groups of subjects are enrolled in the study:
  * patients with a mental disorder
  * relatives of patients included
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Subject suffering from (according to DSM IV criteria)
  * bipolar disorder
  * unipolar depression
  * schizophrenia
  * autism spectrum disorder
  Collection of hair follicle cells
  Interventions: Genetic: study of the transmission of genetic variants
- Relatives (Other): Relatives of enrolled patients suffering from psychiatric disorder.
  * test to detect psychiatric disorders
  * blood or saliva sampling for genomic DNA extraction
  * Collection of hair follicle cells
  Interventions: Genetic: study of the transmission of genetic variants

INTERVENTIONS:
Genetic: study of the transmission of genetic variants — the genetic variants of interest will be investigated by sequencing or genotyping on genomic DNA

SUMMARY:
Genetic analyses conducted on patient with psychiatric disorders assessed at the expert centres resulted in the identific action of genetic variants associated with psychiatric disorders (Courtois, 2020). These data require further genetic and functional analyses. The first objective of this study is to investigate the disease-related inheritance of genetic variants in the families of individuals in whom these variants have been identified. The second objective is to explore the functional consequences of disease-associated genetic variants in patients cells and those of their relatives with and without these variants.

The present project aims to enrich existing biocollections with DNA from blood or saliva from relatives of patients identified with genetic variants. In addition, we wish to collect hair follicules from patients with identified genetic variants of interest and their family members who wish to participate in the study. These hair samples with SNA will be used to dedifferentiate the isolated cells into induced pluripotent stem cells (IPSCs), and then to differentiate them into cells expressing the gene of interest, such as neurons or astrocytes, or into more complex systems, such as brain organoids.

ELIGIBILITY:
Inclusion Criteria:

* For patients:
* Subjects suffering from (according to DSM IV criteria) : Bipolar disorder, Unipolar depression, Schizophrenia, Autism spectrum disorder
* Age over 18 years
* Subject affiliated to the social security system
* Including patients under guardianship, curatorship,
* Patients included in the Fondation FondaMental cohort whose genetic analyses have revealed the need for comparative and functional genetic studies.
* Having signed the consent form

For relatives :

* Age over 18 years
* Relative of patient included in the Fondattion FondaMental cohort
* Including relative under guardianship, curatorship
* Having signed the consent
* Affiliated to social security

Exclusion Criteria:

* For all subjects:
* Any condition that, in the opinion of the investigator, would make the subject's participation in the study undesirable or that would compromise compliance with the protocol
* Persons deprived of liberty
* Inability to understand French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Measure of the probability of having a psychiatric disorder given the presence of the genetic variant studied. | through study completion, an average of 5 years
  Test for psychiatric disorders Study of the genetic variant of interest by sequencing or genotyping on genomic DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Leboyer, MD PhD, Study Chair — Fondation FondaMental; Stephane JAMAIN, PhD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hopital Albert Chenevier, Créteil, France

IPD SHARING:
Plan to Share IPD: No